CLINICAL TRIAL: NCT05484245
Title: Sonography-guided Resection of Brain Mass Lesions: a Prospective, Single Arm Clinical Trial
Brief Title: Sonography-guided Resection of Brain Mass Lesions
Acronym: SOMALI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Principal Investigator, Sklifosovsky Institute of Emergency Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9g
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tumor, Brain; Arteriovenous Malformations; Cavernoma; Intracerebral Hematoma
Keywords: intraoperative sonography; intraoperative ultrasound; brain tumor; cavernoma; arteriovenous malformation; intracerebral hematoma
MeSH Terms: conditions — Brain Neoplasms; Arteriovenous Malformations; Hemangioma, Capillary; Cerebral Hemorrhage | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery (Experimental): Ultrasound-guided resection of brain tumors, vascular malformations and hematomas
  Interventions: Device: Sonography

INTERVENTIONS:
Device: Sonography — Surgeon detects brain mass lesion and assesses extent of it's resection with sonography

SUMMARY:
Objective of the study is to determine possibilities of intraoperative sonography in detecting of various brain mass lesions, assessing extent of their resection and define indications to use ultrasound-guided needle or ultrasound wire-guided port.

DETAILED DESCRIPTION:
Intraoperative sonography is usially used in neurooncology to detect brain tumors and exclude their remnants. A few studies describe it's usage while removing hematomas or vascular malformations. Ultrasound is the only method allowing to observe brain tissue in real time. It is chip and doesn't violate surgical workflow. Main disadvantages of sonography are lengthy learning curve and poorer image quality compared to magnetic resonance imaging. Novel acoustic coupling fluid, contrast-enhanced ultrasound and elastography expanded it's effectiveness. Meanwhile problems of locating of isoechogenic lesions with poor margins and elimination of artefacts are steel actual.

Objective of the study is to determine possibilities of intraoperative sonography in detecting of various brain mass lesions, assessing extent of their resection and define indications to use ultrasound-guided needle or ultrasound wire-guided port.

A surgeon will intraoperatively locate mass lesion and assess extent of it's resection with sonography. Ultrasound scanning will be performed through the same surgical approach or at a distance through enlarged craniotomy, periodically or permanently. To facilitate approach to subcortical and deep small mass lesions ultrasound-guided needle or ultrasound wire-guided port will be used.

ELIGIBILITY:
Inclusion Criteria:

* all intracranial tumors
* cavernomas
* arteriovenous malformations
* spontaneous (non-traumatic) intracerebral hemorrhages
* traumatic intracerebral hemorrhages
* supratentorial localization
* newly diagnosed
* age 18-100 years
* stable hemodynamics

Exclusion Criteria:

* rapid cerebral dislocation
* previously performed brain radiotherapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound features of various brain mass lesions in Mair scale (in grades) | Intraoperatively
  Assessment of target visibility, echogenicity, homogeneity and border demarcation in sonography and their comparison to preoperative computed tomography and magnetic resonance imaging

SECONDARY OUTCOMES:
Sensitivity of intraoperative sonography to detect mass lesion compared to preoperative magnetic resonance imaging or computed tomography (in percents) | Intraoperatively
  Sensitivity = true detection of mass lesion / (true detection of mass lesion + inability to detect mass lesion) x 100
Sensitivity of intraoperative sonography to detect residual mass lesion compared to postoperative magnetic resonance imaging or computed tomography (in percents) | Within 48 hours after surgery
  Sensitivity = true detection of residual mass lesion / (true detection of residual mass lesion + inability to detect residual mass lesion) x 100
Specificity of intraoperative sonography to detect residual mass lesions compared to postoperative magnetic resonance imaging or computed tomography (in percents) | Within 48 hours after surgery
  Specificity = true absence of residual mass lesion / (true absence of residual mass lesion + false detection of residual mass lesion) x 100
Positive predictive value of intraoperative sonography to detect residual mass lesions compared to postoperative magnetic resonance imaging or computed tomography (in percents) | Within 48 hours after surgery
  Positive predictive value = true detection of residual mass lesion / (true detection of residual mass lesion + false detection of residual mass lesion) x 100
Negative predictive value of intraoperative sonography to detect residual mass lesions compared to postoperative magnetic resonance imaging or computed tomography (in percents) | Within 48 hours after surgery
  Negative predictive value = true absence of residual mass lesion / (true absence of residual mass lesion + inability to detect residual mass lesion) x 100
Accuracy of intraoperative sonography to detect residual mass lesions compared to postoperative magnetic resonance imaging or computed tomography (in percents) | Within 48 hours after surgery
  Accuracy = (true detection of residual mass lesion + true absence of residual mass lesion) / (true detection of residual mass lesion + true absence of residual mass lesion + false detection of residual mass lesion + inability to detect residual mass lesion) x 100
Duration of mass lesion removal (in minutes) | Intraoperatively
  How long did in take to remove mass lesion from starting of it's dissection till final evacuation
Extent of resection (in percents) | Within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100
Differentiation between artefacts and residual lesion (Yes or No) | Intraoperatively
  Possibility of ultrasound differentiation between artefacts and residual lesion
Duration of approach to mass lesion using ultrasound-guided needle or ultrasound wire-guided port (in minutes) | Intraoperatively
  Only for subcortical or deep-seated mass lesions. How long did in take to reach margin of mass lesion after dural incision using ultrasound-guided needle or ultrasound wire-guided port
Karnofsky performance status (in percents) | Within 10 days after surgery
  Assessment of patients' possibilities to self-service in Karnofsky Performance Status scale
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No